CLINICAL TRIAL: NCT02355041
Title: Pilot Meal Replacement-Based Diet Effectiveness Study
Brief Title: Meal Replacement Study
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The PI changed institutions
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 14-1212
Record Dates: First submitted 2015-01-30; First posted 2015-02-04 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Obesity
Keywords: diet; body weight; eating; meal replacement
MeSH Terms: conditions — Obesity; Body Weight

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Meal Replacement-based Weight Loss Diet (Experimental): Experimental participants will be instructed to replace 2 meals per day with a PROBAR meal replacement and consume a dinner under 1000 calories or a dinner under 800 calories and a 200 calorie snack for 90 days. No further nutritional advice or education shall be provided.
  Interventions: Behavioral: Meal Replacement-based Weight Loss Diet
- Educational Video (Active Comparator): Control participants will view "The Weight of the World," a 51 min documentary focusing on the topics of obesity and healthy living. Via information presented by medical professionals and lifestyle experts, this film delves into issues related to preventing and combating obesity through healthy lifestyle changes. Major topics include the importance of healthy eating and exercise behaviors and the changes that can be made by communities to reshape our lifestyles. Potential community changes are further addressed with respect to schools by presenting particularly successful programs that have been implemented in some schools. Participants will stream it free on the web.
  Interventions: Behavioral: Educational Video

INTERVENTIONS:
Behavioral: Meal Replacement-based Weight Loss Diet
  Arms: Meal Replacement-based Weight Loss Diet
Behavioral: Educational Video — Via information presented by medical professionals and lifestyle experts, this film delves into issues related to preventing and combating obesity through healthy lifestyle changes. Major topics include the importance of healthy eating and exercise behaviors and the changes that can be made by communities to reshape our lifestyles. Potential community changes are further addressed with respect to schools by presenting particularly successful programs that have been implemented in some schools. Participants will stream it free on the web.
  Arms: Educational Video

SUMMARY:
Adolescent obesity is associated with a number of serious health conditions and most obese adolescents become obese adults. Despite this fact, very few adolescent health centers offer clinical weight loss programs. This is likely because most weight loss programs require extensive resources and are not covered by most health insurance policies. However, this is expected to change since the American Medical Association's recent decision to recognize obesity as a disease. Therefore, it is important to identify simple and effective nonsurgical programs for weight loss, which can be used in adolescent health centers. The investigators are proposing to show that a meal replacement based diet program will be effective in reducing body mass index (weight adjusted for height). In this pilot study, 90 adolescents will either participate in a meal replacement based weight loss program or watch an educational video. Body mass index and body fat will be recorded over time to see if adolescents participating in the meal replacement program lose more weight than those who do not participate in this program.

In order to address this objective, the investigators will assess group differences in body mass index (BMI; kg/m2), body composition (% body fat), eating disorder symptoms and psychological/behavioral variables.

DETAILED DESCRIPTION:
Obesity is a risk factor for a number of serious medical comorbidities and is second only to smoking as the leading cause of preventable death in the US. Further, estimates of the costs associated with overweight and obesity have topped $200 billion annually. The numbers are particularly alarming for adolescents, in whom the rate of obesity has risen at 2-3 times as quickly as in adults. Despite the urgent need, very few clinical centers offer obesity treatment due to the resource-intensive nature of most interventions and the fact that behavioral obesity interventions have rarely been reimbursed by 3rd party payers. Following the American Medical Association's recent decision to recognize obesity as a disease and establish ICD-10-CM Diagnosis Codes (e.g., E66.0), however, there is increasing pressure for 3rd party payers to reimburse for effective obesity interventions. Thus, it is critical to identify effective treatment options that can be implemented in medical centers. Prior research has shown meal replacement-based diets to be more effective than typical "lifestyle-change" diet programs, both in terms of weight loss and, more importantly, weight loss maintenance. Evidence also suggests that solid meal replacements (e.g., bars) show greater effectiveness than liquid meal replacements (e.g., shakes). Finally, greater effectiveness is seen with meal replacements that are higher vs. lower in protein. Importantly, these interventions show high rates of effectiveness even in the absence of nutritional counseling, suggesting that a solid meal-replacement based diet program that is relatively high in protein could be highly effective and easily implemented in clinical settings. In this pilot study, 90 adolescents will be randomized to either a meal replacement-based diet (experimental) group or an educational video (comparison) group.

All recruitment and study procedures will take place at the Mount Sinai Adolescent Health Center (MSAHC). The MSAHC is the largest adolescent-specific, integrated, primary care facility in the U.S., and is a unique model that integrates medical, sexual, reproductive, mental health and health education services. MSAHC provides inner-city youth ages 10-24 who are predominately youth of color high quality, comprehensive, easily accessed, free services. Flyers will be posted in the clinic of the Mount Sinai Adolescent Health Center.

At the baseline assessment following recruitment, participants will provide informed consent and complete a structured interview conducted by research staff to more formally assess eating patterns and eating disorders symptomatology. Assessors will conduct interviews at the MSAHC on an individual basis. If a patient meets criteria for an eating disorder, s/he will be referred to treatment. Participants will be randomly assigned to one of two groups using the coin flipper function available at www.random.org. All files will be password protected to prevent unauthorized access of data.

ELIGIBILITY:
Inclusion Criteria:

* Patient at Mount Sinai Adolescent Health Center
* 18-24 years old
* Obese (BMI at or above the 95th percentile for patients ≤ 20 y.o and BMI ≥ 30 for patients ≥21 y.o.)

Exclusion Criteria:

* Not a patient at Mount Sinai Adolescent Health Center
* Current eating disorder (anorexia nervosa, bulimia nervosa or binge eating disorder)
* Girls who are pregnant or planning to become pregnant. A participant who becomes pregnant during the study will be terminated from the study.
* Patients with diabetes
* Individuals with active psychiatric or substance use disorders
* Individuals who are allergic to tree nuts, peanuts, milk, eggs, wheat, and sesame.
* Normal weight or overweight patients (< 95th percentile)

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | up to 12 months
  - Body mass index (BMI; kg/m2). Height will be measured to the nearest millimeter using a direct reading stadiometer. Weight will be assessed to the nearest 0.1 kg using a digital scale (Tanita TBF-300A) with participants wearing light clothing without shoes or coats.

SECONDARY OUTCOMES:
Body Fat as measured by Bioelectrical impedance analysis (BIA) | up to 12 months
  Bioelectrical impedance analysis (BIA) using the Tanita TBF-300A Body Composition Analyzer to assess % body fat to maximize sensitivity to predict increases in body fat and obesity onset.
Eating Disorder symptoms as measured by the Eating Disorder Diagnostic Scale | up to 12 months
  The Eating Disorder Diagnostic Scale for screening eating pathology
Body Dissatisfaction as measured by an adapted form of the Satisfaction and Dissatisfaction with Body Parts Scale | up to 12 months
  an adapted form of the Satisfaction and Dissatisfaction with Body Parts Scale to assess body satisfaction. It asks respondents to rate their level of satisfaction with nine body parts on 6-point scales ranging from "extremely satisfied" to "extremely dissatisfied."
Depressive symptoms as measured by the 21-item Beck Depression Inventory | up to 12 months
  The 21-item Beck Depression Inventory to assess depressive symptoms
Emotional Eating as measured by the Emotional Eating scale | up to 12 months
  The Emotional Eating scale from the Dutch Eating Behavior Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Ochner, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai